CLINICAL TRIAL: NCT05193838
Title: Effect of Allopurinol on Left Ventricular Function in Children With Dilated Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Seif-elnasr Mohamed, principal investigator, Assiut University
Other Study IDs: Allopurinol
Record Dates: First submitted 2021-11-26; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Allopurinol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allopurinol: we plan to follow up effect of Allopurinol on left ventricular function in children with dilated cardiomyopathy for 6 months
  Interventions: Drug: Allopurinol Tablet

INTERVENTIONS:
Drug: Allopurinol Tablet — examined patients with dilated cardiomyopathy will receive allopurinol for 6 months

SUMMARY:
The aim of this study is to detect effect of allopurinol supplementation in pediatric patients with dilated cardiomyopathy.

DETAILED DESCRIPTION:
DCM as a serious cardiac disorder in which structural or functional abnormalities of the heart muscle can lead to substantial morbidity and mortality owing to complications such as heart failure and arrhythmia Among patients with heart failure (HF), elevated serum uric acid levels and increased oxidative stress have been associated with increased mortality, implicating xanthine oxidase as a possible therapeutic target Xanthine oxidase (XO), a superoxide-generating enzyme, is up regulated in animals (6,7) and in humans with heart failure. Acute administration of the XO inhibitor allopurinol improves the mechanical efficiency of the failing heart ), whereas oxygen consumption paradoxically decreases. Direct XO inhibition in cardiac muscle leads to increased force generation by the myofilaments at any given level of activator calcium(10).

Allopurinol, an inhibitor of xanthine oxidase, may be a novel therapeutic agent for HF. Allopurinol reduces uric acid levels, prevents acute gout, and acts as an anti oxidant, which could be beneficial among HF patients(5)

ELIGIBILITY:
Inclusion Criteria:

1 - children (1-16) year's age with impaired left ventricular systolic function due to dilated cardiomyopathy, who attend pediatric cardiology unit 2-children attend to pediatric cardiology out patient clinic in Assiut university children hospital 3-children with no allergic reaction from allopurinol

Exclusion Criteria:

1. children with impaired left ventricular systolic function due to other causes like congenital heart diseases
2. children with acquired heart diseases
3. patients with allergic reaction or contra indicated from Allopurinol

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is a prospective cohort study, it will include 100 patient who attend pediatric cardiology unit or pediatric cardiology outpatient clinic in Assiut university children hospital in Assiut governate, Egypt
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
difference of echocardiography parameters and ejection fraction between DCM patients taking Allopurinol and patients not taking | 6 months
  follow up of improvement of ejection fraction by echocardiography

REFERENCES:
- [Background] Maron BJ, Towbin JA, Thiene G, Antzelevitch C, Corrado D, Arnett D, Moss AJ, Seidman CE, Young JB; American Heart Association; Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; Council on Epidemiology and Prevention. Contemporary definitions and classification of the cardiomyopathies: an American Heart Association Scientific Statement from the Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; and Council on Epidemiology and Prevention. Circulation. 2006 Apr 11;113(14):1807-16. doi: 10.1161/CIRCULATIONAHA.106.174287. Epub 2006 Mar 27. PMID 16567565